CLINICAL TRIAL: NCT01967901
Title: Impact of a Multidisciplinary Self-care Management Program on Quality of Life, Self-care Behavior, Adherence to the Anti-hypertensive Treatment, Glycemic Control, and Renal Function in Adults Living With Diabetic Kidney Disease
Brief Title: Impact of Multidisciplinary Self-care Management of Diabetic Nephropathy on Quality of Life, Self-care Behavior, Glycemic Control, and Renal Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Collaborators: University of Lausanne (Other); University of Lausanne Hospitals (Other); Leenaards Fondation, Switzerland (Unknown)
Responsible Party: Principal Investigator, Nancy Helou, Lecturer at University of Applied Sciences of Western Switzerland, PhD (c) at the University of Lausanne, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 37319/S-RAD13-07
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic nephropathies; Nursing; Multidisciplinary; Self-care; Quality of Life
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sequence: ABBA A=usual care, B=self-care (Active Comparator): The usual care consists of patients' follow up by their usual nephrologist and endocrinologist or general practitioner.
  Self-care management consists of a the addition of a multidisciplinary self-management program that includes additional home and clinic visits and telephone follow-ups made by the self-care management nurse and clinic visits to the dietician.
  In this sequence, patients will receive the usual care for 3 months. Then, they will cross-over to receive a multidisciplinary self-management for the following 6 months and then cross-over to a 3 months of usual care.
  Interventions: Behavioral: Self-care management program
- Sequence BAAB (Active Comparator): Patients will receive the multidisciplinary self-management program for 3 months. Then, they will cross-over to usual care for the following 6 months and then cross-over to 3 months of multidisciplinary self-management
  Interventions: Behavioral: Self-care management program
- Sequence AABB (Active Comparator): Patients will receive the usual care for two periods of three months, then they will cross-over to a period of 6 months of a multidisciplinary self-management
  Interventions: Behavioral: Self-care management program
- Sequence BBAA (Active Comparator): Patients will receive the multidisciplinary self-management for two periods of three months, then they will cross-over to a period of 6 months of usual care.
  Interventions: Behavioral: Self-care management program

INTERVENTIONS:
Behavioral: Self-care management program — The self-care management consists of the usual care with an additional multidisciplinary self-management program that includes additional home and clinic visits and telephone follow-ups made by the self-care management nurse and clinic visits to the dietician.

SUMMARY:
Diabetic Kidney Disease (DKD) is becoming a global health concern that affects largely the elderly population. Despite advances in pharmacological and management strategies, DKD remain associated with high morbidity and mortality. Patients living with such chronic disease, are expected, on daily basis to manage their self-care activities. Patients' non-adherence to the treatment is thought to be the major cause for the poor control and the occurrence of complications. Previous researchers have shown that multidisciplinary management of chronic disease can improve patients' self-care and outcomes. However, none of these programs was centered on self-care and targeted patients with DKD. A multidisciplinary self-care management program could improve the outcomes of patients with DKD, and delay the progression of the disease.

The aim of the study is to investigate the effect of a multidisciplinary self-care management program on self-care behavior, quality of life, medication adherence, glycemic control and renal function, in adults with DKD.

The study will use a cross-over design. 32 adult with DKD, will be randomly recruited from the Vaud University Medical Center, nephrology department and will be enrolled in the program for 12 month. All variables will be measured at baseline, three, six, nine and 12 month. We will measure the patients' self-care behavior, quality of life, adherence to the anti-hypertensive medication taking using, the Revised Summary of Diabetes Self-Care Activities questionnaire, the Audit of Diabetes-Dependent Quality of life questionnaire and the Medication Events Monitoring System. We will assess the patients' glycemic control by measuring the glycated hemoglobin and the renal function by measuring the serum creatinine and the microalbumin creatinine ratio.

The study will clearly show if a multidisciplinary self-care management program will improve the health outcomes of patients with DKD and will allow us to recommend the establishment of such a program.

ELIGIBILITY:
Inclusion Criteria:

* Age eighteen and more
* Clinical diagnoses of diabetes
* Clinical diagnosis of renal disease and an Estimated Glomerular Filtration Rate (eGFR) of less than 60ml/min calculated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD_EPI) formula and /or an Albumin/Creatinine ratio of 30mg/mmol or more.
* Free of cognitive deficit as determined by the recruiting nephrologist based on a normal score on the Short Portable Mental Status Questionnaire.

(The nephrologist will ensure patients' referral or follow-up in the case of a diagnosed cognitive deficit)

* Free of psychomotor skills limitations as determined by the physical examination of the medical doctor recruiting the patient.
* Able to read, write and speak in French

Exclusion Criteria:

* Terminal illness other than chronic kidney disease such as cancer or severe heart failure.
* Planned major surgical procedures.
* Patient on dialysis.
* Patient receiving nursing home care visits for the management of diabetes.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months
  The Quality of life will be measured using the French version of the Audit of Diabetes-Dependent Quality of life (ADDQoL) measure at baseline, at the end of three months of follow-up, at the end of six months of follow-up, at the end of nine months of follow-up, and at the end of twelve months of follow-up.

SECONDARY OUTCOMES:
Self-care | 12 months
  Self-care behavior will be measured using the French translated version of the Revised Summary of Diabetes Self-Care Activities(R-SDSCA)
The adherence to anti-hypertensive medication | 12 months
  The adherence to anti-hypertensive medication taking will be measured using the Medication Events Monitoring system (MEMS)
Blood glucose control | 12 months
  The blood glucose control will be evaluated through the measurement of the glycated hemoglobin HbA1C
Kidney function | 12 months
  The kidney function will be evaluated through the measurement of the serum creatinine, and the microalbumin creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Maya Shaha, PhD, RN, Study Director — University of Lausanne- Faculty of Biology and Medicine, Institut universitaire de formation et de recherche en soins
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Hodson EM, Cooper TE. Altered dietary salt intake for preventing diabetic kidney disease and its progression. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD006763. doi: 10.1002/14651858.CD006763.pub3. PMID 36645291
- [Derived] Helou N, Talhouedec D, Shaha M, Zanchi A. The impact of a multidisciplinary self-care management program on quality of life, self-care, adherence to anti-hypertensive therapy, glycemic control, and renal function in diabetic kidney disease: A Cross-over Study Protocol. BMC Nephrol. 2016 Jul 19;17(1):88. doi: 10.1186/s12882-016-0279-6. PMID 27430216